CLINICAL TRIAL: NCT04654065
Title: An Open-label, Single-dose Clinical Study to Evaluate Oral Mucosa Absorption of IN-C004 in Healthy Volunteers
Brief Title: Study to Evaluate Oral Mucosa Absorption of IN-C004 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IN_KOD_101
Record Dates: First submitted 2020-11-29; First posted 2020-12-04 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IN-C004 (Experimental): IN-C004
  Interventions: Drug: IN-C004

INTERVENTIONS:
Drug: IN-C004 — One time dose of IN-C004 taken orally.

SUMMARY:
To evaluate whether IN-C004 absorbs oral mucosa in healthy volunteers.

DETAILED DESCRIPTION:
An Open-label, Single-dose Clinical Study

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥19.0 kg/m2 and ≤27.0 kg/m2 with a body weight ≥ 45 kg at screening.

Exclusion Criteria:

* History or evidence of clinically significant disease
* History of drug/alcohol abuse
* Participated in other studies and received investigational products within 6 months prior to the first study dose.
* Not able to use a medically acceptable contraceptive method throughout the study.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
AUCt of tegoprazan | pre-dose(0 hour), 0.08, 0.17, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 2 hours
  Area under the plasma concentration-time curve of tegoprazan
Cmax of tegoprazan | pre-dose(0 hour), 0.08, 0.17, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 2 hours
  Maximum Plasma Concentration at Steady State of tegoprazan
Tmax of tegoprazan | pre-dose(0 hour), 0.08, 0.17, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 2 hours
  Time to reach Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea